CLINICAL TRIAL: NCT01760733
Title: Improved Selection of Elderly (> 65 Years) for Kidney Transplantation
Acronym: QUESTION65
Status: Active, not recruiting | Type: Observational
Sponsor: Sykehuset Telemark (Other Government)
Collaborators: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Kristian Heldal, Consultant nephrologist, PhD, MHA, Sykehuset Telemark
Other Study IDs: STHF 81.25
Record Dates: First submitted 2012-12-17; First posted 2013-01-04 (Estimated); Results first posted 2020-04-24 (Actual); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Quality of Life; End Stage Renal Disease; End Stage Renal Failure on Dialysis
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Kidney transplantation has been shown to provide improved survival even in patients older than 70 years of age. The purpose of the study is to determine whether kidney transplantation provides any improvement of health related quality of life (HRQOL) in patients over the age of 65 years. HRQOL wil be monitored using the Kidney Disease and Quality of Life (KDQOL-SF)form. Patients will be recruited at the time of acceptance to the Norwegian transplant wait list and followed every 6 months until transplantation. Thereafter a new form will be completed after 10 weeks post transplant, 6 months, 1 year, 3 years and 5 years. In addition the study will explore the transplant candidates expectations in a qualitative study design and explore the relationship between pre-transplant comorbidity, HRQOL and survival.

DETAILED DESCRIPTION:
Aim 1:

Evaluate the HRQoL longitudinally from time of wait listing and until 1 year after kidney transplantation among kidney transplant candidates older than 65 years of age.

Data collection The HRQoL will be monitored in a prospective, longitudinal study (QUESTION65). A minimum of 200 patients will be included and the inclusion period is estimated to 2-3 years. All patients give informed consent when entering the study. In addition, all patients have signed an informed consent when included in the Norwegian Renal Registry which allows the use of unidentified data from the registry in research protocols.

HRQoL will be assessed using the Kidney Disease Quality of Life Short Form (KDQOL-SF-36) health Survey. This survey consists of two parts, a generic and disease specific part. The same questionnaire is used before and after transplantation. For improved evaluation of HRQoL data on response shift will be captured through questions related to personal preferences, values and internal standards. The result gathered will also be compared with data from an age matched Norwegian cohort.

All patients over the age of 65 who are accepted for the kidney transplantation waiting list or living donor transplantation will receive an invitation to be included in the study. A new form will be distributed to included patients with intervals of six months until they are transplanted, permanently removed from the transplant waiting list or until death. Patients who are transplanted will receive a form at discharge from Oslo University Hospital, Rikshospitalet (10 weeks after transplantation), after six months and at one year.

Aim 2:

Explore the expectations of older kidney transplant candidates prior to transplantation and one year after transplantation.

Data Collection:

For the qualitative evaluation, 15-20 patients in dialysis will be included and a qualitative individual in-depth interview will be performed approximately one month after baseline HRQoL and repeated one year after transplantation. Selection will be made according to age and gender. Inclusion will continue until saturation is reached. Convenient variation and broadness in information will be secured in the sample. To secure shared decision making, patients will be invited to discuss the interview guide and design of the qualitative evaluation. Furthermore, the interview guide will be tested in a pilot study. An interview-manual will be used. We believe the results from the qualitative interviews also can be used to gain an improved understanding of the answers in the survey.

Aim 3:

Investigate the relationship between pre-transplant comorbidity, described by the Liu comorbidity index and post-operative complications, post-transplant 1 year survival and HRQoL.

Data collection From 2012 we have included pre-transplant data according to the Liu comorbidity index as part of the routine work up of candidates for kidney transplantation. Complete data describing patient and transplant characteristics, including the Liu comorbidity index will be extracted from the Norwegian Renal Registry. These data will only be used as explanatory variables for the outcome of HRQoL/survival and are not reported as separate outcomes. In addition post-transplant morbidity and mortality will be extracted from the Norwegian Renal Registry. The data will be exported from the registry without any identification except from a patient number.

In case of missing data from the registry, data will be retrieved from the patient records at Oslo University Hospital, Rikshospitalet. The key necessary for identification will be stored at the registry.

Aim 4 Health economic evaluation. In this sub-study, we will use data from the Short Form 36 (SF36) part of the KDQOL-SF questionnaire to calculate Quality Adjusted Life Years (QALY). Costs will be estimated for each patients using data from their hospital records.

ELIGIBILITY:
Inclusion Criteria:

* End stage renal disease listed for transplantation
* Age > 65 years

Exclusion Criteria:

* Not able to fulfill the HRQOL form

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients older than 65 years listed for kidney transplantation on the Norwegian transplant wait list
Sampling Method: Non-Probability Sample
Enrollment: 289 (Actual)
Dates: Start 2012-12; Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Kristian Heldal, MD, PhD, Principal Investigator — Sykehuset Telemark
Locations (1):
- Oslo University Hospital, Rikshospitalet, Section of Nephrology, Oslo, Norway

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Lonning K, Midtvedt K, Heldal K, Andersen MH. Older kidney transplantation candidates' expectations of improvement in life and health following kidney transplantation: semistructured interviews with enlisted dialysis patients aged 65 years and older. BMJ Open. 2018 Jun 22;8(6):e021275. doi: 10.1136/bmjopen-2017-021275. PMID 29934388
- [Result] Lonning K, Heldal K, Bernklev T, Brunborg C, Andersen MH, von der Lippe N, Reisaeter AV, Line PD, Hartmann A, Midtvedt K. Improved Health-Related Quality of Life in Older Kidney Recipients 1 Year After Transplantation. Transplant Direct. 2018 Mar 1;4(4):e351. doi: 10.1097/TXD.0000000000000770. eCollection 2018 Apr. PMID 29707622
- [Result] Lonning K, Midtvedt K, Bernklev T, Brunborg C, Andersen MH, von der Lippe N, Reisaeter AV, Line PD, Hartmann A, Heldal K. Changes in health-related quality of life in older candidates waiting for kidney transplantation. Nephrology (Carlton). 2018 Oct;23(10):948-956. doi: 10.1111/nep.13117. PMID 28734131

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All patients 65 years and older who were accepted on the Norwegian kidney transplantation waiting list between January 1st 2013 and November 30th 2016 were invited to participate (n = 437). 289 were included, reasons for exclusion were reluctant to participate ( n = 21), not meeting inclusion criteria (n = 21) and not responding (n = 105).
Groups:
- Patients Accepted for the Transplant Waiting List: Patients accepted for the kidney transplantation waiting list at Oslo University Hospital between Jan 1 2013 and Nov 30 2016 were included and followed from time of acceptance and up to 10 years after transplantation
Period: Waiting List
Arm/Group | Patients Accepted for the Transplant Waiting List
Started | 289 (All patients included started in the waiting list group.)
Completed | 217 (217 patients have been transplanted)
Not Completed | 72
Not completed — Death | 18
Not completed — Removed from waiting list | 41
Not completed — Not received a transplant yet | 13
Period: Transplanted
Arm/Group | Patients Accepted for the Transplant Waiting List
Started (By Sept 15 2019, 217 patients have received a kidney transplant) | 217
Completed (By Sept 15 2019, 8 patients have died after kidney transplantation) | 0
Not Completed | 217
Not completed — Not reached 10 years post transplant | 184
Not completed — Death | 26
Not completed — Graft loss | 7

BASELINE CHARACTERISTICS:
Population: Patients older than 65 year accepted for KTx
Groups:
- Waiting List: Patients on the waiting list for transplantation
Arm/Group | Waiting List
Number analyzed (Participants) | 289
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 289
Age, Continuous [Mean (Full Range); unit: years] | 70.6 [64.8 to 82.2]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 93
  Male | 196
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Norway | 289
Health Related Quality of Life scores (KDQOL-SF) [Mean (Standard Deviation); unit: scores on a scale SF-36 general health] — The KDQOL-SF questionnaire was distributed by mail to all included patients at baseline. The questionnaire consist of a generic part (SF-36, 8 domains, and a disease specific part (KDQOL, 11 domains). The scores of all dimensions ranging between 0 and 100 with higher scores indicating better outcomes, were used separately in further analyses. The patients completed the questionnaire without any assistance from health personnel.
  In this report we only report the scores for the dimension general health (GH)
  scores on a scale SF-36 general health | 49.9 (22.3)

OUTCOME MEASURES:

1. Primary Outcome: Changes in Short-term (One Year) Health Related Quality of Life, Measured by the KDQOL-SF Questionnaire
Description: Longitudinally monitoring of health related quality of life (HRQOL) by the Kidney Disease and Quality of Life Short Form (KDQOL-SF) questionnaire from listing for transplantation and up to one year post transplantation. The KDQOL-SF scores are organized in 18 dimensions and the Scores for each Dimension are reported within the range 0-100, higher scores indicate better Health related quality of life. Scores are obtained at baseline and every six months while patients were on the waiting list are performed. In addition scores are obtained obtained at two, six and twelve months after transplantation. Comparisons between last score obtained on the waiting list and score at twelve months after transplantation are performed. The results are reported as absolute values and changes from baseline/last score before transplantation and the scores at one year post transplant.
Time Frame: Change in health related quality of life from baseline to one year after transplantation
Population: Changes in SF-36 score for the dimension "general health" (GH) of the KDQOL-SF between baseline and one year after transplantation
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Waitlist: Patients on the waiting list for transplantation
- Transplanted: Patients who have received a transplant
Arm/Group | Waitlist | Transplanted
Number analyzed (Participants) | 289 | 217
score on a scale | 49.5 (22.3) | 68 (22)

2. Primary Outcome: Health Economic Analyses
Description: Quality Adjusted Life Years (QALY) are calculated based on Short Form-6D extracted from the SF-36 part of the KDQOL survey while patients were on the waiting list and after transplantation. QALYs are compared between the waiting list and up to three years after transplantation. Costs will be calculated based on information from the patients records and cost/QALY will be compared for the two periods
Time Frame: From baseline to three years post transplant
Reporting Status: Not Posted, anticipated posting 2021-06

3. Primary Outcome: Survival
Description: Patient survival on the waiting list and after transplantation will be calculated and compared using the Kaplan Meier method and a Cox regression analysis with a time dependent variable.
Time Frame: From baseline/last score before transplantation to transplantation/up to ten years post transplant
Reporting Status: Not Posted, anticipated posting 2022-12

4. Primary Outcome: Changes in Intermediate Term (Three Years) Health Related Quality of Life, Measured by the KDQOL-SF Questionnaire
Description: Longitudinally monitoring of health related quality of life (HRQOL) by the Kidney Disease and Quality of Life Short Form (KDQOL-SF) questionnaire from listing for transplantation and up to three years post transplantation. The KDQOL-SF scores are organized in 18 dimensions and the Scores for each Dimension are reported within the range 0-100, higher scores indicate better Health related quality of life. Scores obtained at baseline and every six months while patients were on the waiting list. In addition scores are obtained at two, six, twelve months and at three years after transplantation. For this outcome, comparison between last score obtained on the waiting list and the score at three years post transplant is performed. The results are reported as absolute values and changes from baseline/last score before transplantation and the score at three years post transplant.
Time Frame: From baseline to three years post transplant
Reporting Status: Not Posted, anticipated posting 2020-12

5. Primary Outcome: Changes in Long Term (5-10 Years) Health Related Quality of Life, Measured by the KDQOL-SF Questionnaire
Description: Longitudinally monitoring of health related quality of life (HRQOL) by the Kidney Disease and Quality of Life Short Form (KDQOL-SF) questionnaire from listing for transplantation and up to three years post transplantation. The KDQOL-SF scores are organized in 18 dimensions and the Scores for each Dimension are reported within the range 0-100, higher scores indicate better Health related quality of life. Scores obtained at baseline and every six months while patients were on the waiting list. In addition, scores are obtained at two, six, twelve months and at three years after transplantation. For this outcome, comparisons between last score obtained on the waiting list and the score at five and ten years post transplant are performed. The results are reported as absolute values and changes from baseline/last score before transplantation and the score at five and ten years post transplant.
Time Frame: From last score before transplantation to ten years post transplant
Reporting Status: Not Posted, anticipated posting 2025-12

6. Secondary Outcome: Associations Between Pre-transplant Patient and Transplant Characteristics and Intermediate Term (Three Years) Change in HRQoL
Description: Demographic, medical and transplant characteristics were included in multivariable regression models to analyze any associations between these variables and any change in HRQoL described as KDQOL-SF scores between last score before transplantation and three years post transplantation
Time Frame: From last score before transplantation to three years post transplant
Reporting Status: Not Posted, anticipated posting 2021-06

7. Secondary Outcome: Associations Between Pre-transplant HRQoL/Comorbidity and Post Transplant Survival
Description: Any associations between pre-transplant HRQoL/comorbidity and post transplant survival will be investigated using multivariable cox regression models.
Time Frame: From transplantation and up to ten years post tx
Reporting Status: Not Posted, anticipated posting 2022-12

ADVERSE EVENTS:
Time Frame: This is an observational study describing HRQoL among elderly Kidney Transplant candidates, longitudinally before and after KTx. No experimental interventions are performed and consequently adverse advents other than death, graft loss and being removed from the waiting list are not collected. Data are reported continuously from the clinicians to the Norwegian Renal Registry and exported to the study database. We search the registry every month and update our study database accordingly.
Description: The term serious adverse event describes number of patients who are removed from the transplantation waiting list because of medical reasons and patients with graft loss after transplantation.
  All cause mortality is reported from both patients on the waiting list and those who have received a transplant.
Groups:
- Question 65: Patients on the waiting list for transplantation - 5 years post KTx Observational study
Arm/Group | Question 65
All-Cause Mortality (participants affected / at risk) | 44/289
Serious Adverse Events (participants affected / at risk) | 48/289
Other Adverse Events (participants affected / at risk) | 0/289
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Question 65 (N=289)
Graft loss (Renal and urinary disorders) | 7/217 (7) — Loss of function of kidney transplant
Removed from the transplantation wait-list (General disorders) | 41 (41) — Patients who are removed from the transplantation waiting list because of medical conditions making the ineligible for the procedure

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-05): https://cdn.clinicaltrials.gov/large-docs/33/NCT01760733/Prot_SAP_000.pdf